CLINICAL TRIAL: NCT00592800
Title: Evaluation of the Understanding of Probability in Children
Brief Title: Understanding Probability in Children
Status: Terminated | Type: Observational
Why Stopped: Lack of study funding & resources
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Arjunan Ganesh, MBBS, The Children's Hospital of Philadelphia
Other Study IDs: 2007-1-5125
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Understanding Probability
Keywords: statistics; probability

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: children between 11 and 13 years of age
- 2: children between 14 to 15 years of age
- 3: children between 16 and 18 years of age

SUMMARY:
To make medical decisions involving pros and cons, one also has to understand probability and percentages. This is a preliminary study to evaluate the ability of children to understand probability and percentages.

DETAILED DESCRIPTION:
The concept of patients making decisions with respect to their health care is well accepted in adult medicine but, the value and importance of decision making in the care of children is not recognized. The major objection raised against allowing children to express their opinions concerning outcomes is that children do not understand probability.

One way of assessing children's ability to understand probability is to test their mathematical knowledge using tests focused on probability and percentage.

We have designed a set of questionnaires with 10 questions each, taken from the US Department of Education's National Assessment of Educational Progress (NAEP). They are divided into 3 different groups (4th, 8th, and 12th grade), based on grade-level. We have also obtained the average percentage of correct-incorrect answers given to these questions by students nationwide, and the scoring system used to assess the student's proficiency level.

In this preliminary study we intend to present this set of 10 mathematical questions to children and to one of their parents.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages 11 to 18 years.
2. Spoken and written English as primary language of both parents and children.
3. Children scheduled to receive anesthesia.
4. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Children with known mental retardation, of any nature.
2. Children who attend schools for children with special needs.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This prospective study will involve one or two encounters with each child and a parent at the Anesthesia Resource Center (ARC) at The Children's Hospital of Philadelphia (CHOP) and the second visit at CHOP during the post-operative phase of recovery prior to discharge from the hospital.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To compare the percentage of children who answer correctly to a set of mathematical questions to verify the ability of children to understand probability and percentages. The results will be compared to those obtained in children nationwide in 2003. | During pre-operative visit.

SECONDARY OUTCOMES:
The secondary objective is to compare the responses between children and parent. | During the pre-operative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Arjunan Ganesh, MBBS, Principal Investigator — Children's Hospital of Philadelphia